CLINICAL TRIAL: NCT00165919
Title: Immunologic Determinants of Hepatitis C Virus Infection Resolution or Persistence
Brief Title: Immune Response to Hepatitis C Virus
Status: Withdrawn | Type: Observational
Why Stopped: Not a clinical trial; human specimens from treatment site for basic research.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Arash Grakoui PhD, Associate Professor, Emory University
Other Study IDs: 1358-2004
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Hepatitis C; HIV Infections
Keywords: Hepatitis C; HIV; Immunopathogenesis; HIV-1
MeSH Terms: conditions — Hepatitis C; HIV Infections | interventions — Laboratories

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HCV+: No group or cohort; not a clinical trial
  Interventions: Other: None. Not a clinical trial. Specimens taken for basic research in laboratory.

INTERVENTIONS:
Other: None. Not a clinical trial. Specimens taken for basic research in laboratory.

SUMMARY:
The purpose of the study is to investigate the immune response to hepatitis C virus to determine why some people clear the virus and others develop chronic infection. Changes in immune response once hepatitis C therapy is begun will also be examined. If patients are also HIV+, the effect of antiretroviral therapy on the recovery of hepatitis C immunity will be investigated.

DETAILED DESCRIPTION:
We will analyze the peripheral (blood) and intrahepatic (liver) immune response in hepatitis C infection in patients with clear hepatitis C infection and those who develop chronic infection. We hope to determine immune responses that are important for eliminating the infection. Currently, the treatments for hepatitis C are not effective for everyone. For those patients enrolled who begin hepatitis C treatment, we will evaluate the immune system of people who respond compared to those who do not respond. If the patient is HIV positive, the change in hepatitis C immune response once various HIV medicines (antiretrovirals) are started will also be examined. Any treatment for hepatitis C or HIV will be determined by the patient's primary physician and will not be affected by enrollment in the study.

Blood samples of ~70 cc will be obtained no more than once per week. Patients who begin hepatitis C therapy or antiretroviral therapy if HIV coinfected will provide serial specimens for examination. Patients who undergo liver biopsy as a part of their routine hepatitis care will provide a sample for further studies of the immune response to see if it is different in the liver compared to the blood.

ELIGIBILITY:
This is not a clinical trial.

Inclusion Criteria

* HCV infected and uninfected (controls)
* Women
* Minorities

Exclusion Criteria

* Children
* Individuals who cannot or will not provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is not a clinical trial, but rather a basic science study using blinded human specimens.
  Individuals with HCV infection will be identified for enrollment into our study by our clinical collaborators at the Crawford Long Infectious Diseases Clinic-Emory University. Control individuals with no prior exposure to HCV will be identified and enrolled both from the Crawford Long clinics and from the investigative donor pool at the Emory Vaccine Center. Inclusion in the current study will be limited to individuals with HCV genotype 1 infection as well as uninfected normal controls as determined by antibody and viral load measurements.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-09; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
This is NOT a clinical trial; thus no outcomes. Specimens from human subjects taken at clinical site and sent unidentified to laboratory for assays. | no outcomes measured

SECONDARY OUTCOMES:
This is NOT a clinical trial; thus no outcomes. Specimens from human subjects taken at clinical site and sent unidentified to laboratory for assays. | no outcomes to measure

OTHER OUTCOMES:
This is NOT a clinical trial; thus no outcomes. Specimens from human subjects taken at clinical site and sent unidentified to laboratory for assays. | no outcomes measured

CONTACTS AND LOCATIONS:
Overall Officials: Arash Grakoui, Ph.D., Principal Investigator — Emory University

REFERENCES:
- [Background] Spellberg B, Edwards JE Jr. Type 1/Type 2 immunity in infectious diseases. Clin Infect Dis. 2001 Jan;32(1):76-102. doi: 10.1086/317537. Epub 2000 Dec 15. PMID 11118387